CLINICAL TRIAL: NCT04116125
Title: A Randomized Trial of Sentinel Lymph Node Biopsy vs Radiotherapy Alone After Neoadjuvant Chemotherapy in Patients Undergoing Breast Conserving Surgery With cT1-3N1, ycN0 Breast Cancer
Brief Title: Omitting Biopsy of SEntinel Lymph Node With Radiation After Neoadjuvant Chemotherapy in Breast Cancer (OBSERB) Trial
Acronym: OBSERB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Collaborators: Korean Breast Cancer Study Group (Other)
Responsible Party: Principal Investigator, JeeYeon Lee, Clinical professor, Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-09-023
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Breast Neoplasm Female; Lymphatic Metastasis
Keywords: Breast cancer; cN1, ycN0; Neoadjuvant cheotherapy; Sentinel Lymph Node; Radiotherapy
MeSH Terms: conditions — Lymphatic Metastasis; Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sentinel lymph node biopsy (Placebo Comparator): Perform conventional sentinel lymph biopsy
  Interventions: Procedure: Radiotherapy
- Adjuvant radiation without Sentinel lymph node biopsy (Experimental): Perform radiotherapy instead of sentinel lymph node biopsy
  Interventions: Procedure: Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy — Adjuvant radiotherapy on axillary region

SUMMARY:
The OBSERB study is a multi-center, non-blinded, pragmatic, parallel, randomized controlled trial in which patients with cT1-3N1 and ycN0 breast cancer.

DETAILED DESCRIPTION:
The OBSERB study aims to compare the oncologic outcomes of radiotherapy without sentinel lymph node biopsy versus sentinel lymph node biopsy for the management of breast cancer which showed the cN1 was conversed as ycN0 after neoadjuvant chemotherapy.

To verify whether, the radiotherapy without SLN can be applied, when the cN1 was conversed as ycN0 after neoadjuvant chemotherapy.

To verify whether, the additional treatment decision can be established based on only the biology of primary tumor without the pathologic information of axillary lymph nodes To verify whether, the patients' quality of life can be improved by a less invasive surgical procedure, when the cN1 was conversed as ycN0 after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. women aged > 20 years
2. cT1-3N1M0, primary invasive
3. initially confirmed ALN by fine needle aspiration cytology before neoadjuvant chemotherapy
4. completion of neoadjuvant chemotherapy
5. tumors negative for LN metastasis confirmed by imaging after neoadjuvant chemotherapy

Exclusion Criteria:

1. synchronous distant metastases
2. previous other malignancy
3. bilateral breast cancer
4. previous primary systemic therapy
5. pregnancy or breastfeeding
6. pre-operative radiological evidence of multiple involved or suspicious axillary nodes
7. patient with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Disease free survival including breast, axilla and other organs from medical record

SECONDARY OUTCOMES:
Local recurrence | 5 years
  Ipsilateral breast from medical record
Axillary recurrence | 5 years
  Ipsilateral axillary lymph nodes from medical record
distant recurrence | 5 years
  Other organs except ipsilateral breast and axillary lymph nodes from medical record
distant free survival | 5 years
  No disease on other organs except ipsilateral breast and axillary lymph nodes from medical record
Overall survival | 5 years
  Overall survival from medical record

OTHER OUTCOMES:
Quality of life by questionnaire | 5 years
  Pain, Discomfort, Numbness, Rotation of arm, Lymphedema of arm

IPD SHARING:
Plan to Share IPD: No